CLINICAL TRIAL: NCT05917223
Title: The Impact of Plant-based Protein Blends, With or Without Resistance Exercise, on Skeletal Muscle Protein Synthesis Rates in Older Men and Women
Brief Title: The Impact of Plant-based Blends on Skeletal Muscle Protein Synthesis Rates in Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16408
Record Dates: First submitted 2023-06-11; First posted 2023-06-23 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Nutrition, Healthy
Keywords: Plant-based protein, Protein quality

STUDY DESIGN:
Intervention Model Description: This study is double-blind, placebo-controlled, randomized parallel control trial
Who Masked: Participant, Investigator
Masking Description: This study is double-blind, placebo-controlled, randomized parallel control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Milk protein ingestion (Experimental): Consuming 20 g of Milk Protein dissolved in 350mL of water, one time at the experiment visit
  Interventions: Dietary Supplement: Milk protein ingestion
- Corn protein ingestion (Experimental): Consuming 20 g of Corn protein isolation dissolved in 350mL of water, one time at the experimental visit
  Interventions: Dietary Supplement: Cron protein ingestion
- Corn+Pea protein ingestion (Experimental): Consuming 20 g of Corn+Pea protein isolation dissolved in 350mL of water, one time at the experimental visit
  Interventions: Dietary Supplement: Corn+Pea protein ingestion
- Non-protein, low energy (Experimental): Consuming 20 g of carbohydrate dissolved in 350mL of water, one time at the experimental visit
  Interventions: Dietary Supplement: Non-protein, low energy

INTERVENTIONS:
Dietary Supplement: Milk protein ingestion — It's just an acute intervention, so the participant assigned to the Milk protein ingestion group will consume 20 g of milk protein during infusion protocol.
  Arms: Milk protein ingestion
Dietary Supplement: Cron protein ingestion — It's just an acute intervention, so the participant assigned to the Corn protein ingestion group will consume 20 g of corn protein isolation during infusion protocol.
  Arms: Corn protein ingestion
Dietary Supplement: Corn+Pea protein ingestion — It's just an acute intervention, so the participant assigned to the Corn+Pea protein ingestion group will consume 20 g of Corn+Pea protein isolation during infusion protocol.
  Arms: Corn+Pea protein ingestion
Dietary Supplement: Non-protein, low energy — It's just an acute intervention, so the participant assigned to the Non-protein, low energy group will consume 20 g of carbohydrate during infusion protocol.
  Arms: Non-protein, low energy

SUMMARY:
Lifestyle interventions such as physical activity and dietary habits are the most effective non-pharmacological strategies to combat the loss of muscle mass and the development of mobility limitations with aging. Resistance training (i.e., strengthening exercise) provides a strong stimulus to build muscle mass, and protein provides the essential building blocks. Therefore, an individual's dietary practices can influence the effectiveness of an exercise program - when combined, they work together to increase the muscle-building response. However, not all proteins are equally effective at bringing about muscle growth.

Therefore, the purpose of this study is to investigate the effect of a higher-quality plant-based protein blend with lifting weight on muscle building in older men and women.

DETAILED DESCRIPTION:
Dietary interventions are similarly pertinent in preventing skeletal muscle mass losses with aging. Dietary protein ingestion provides the necessary substrates (i.e., amino acids) essential for skeletal muscle development, health, and, thus, maintenance of muscle mass. Protein ingestion and resistance exercise training (RET) increase muscle protein synthesis (MPS), but when combined, they act synergistically to maximize MPS. Importantly, not all protein sources are equivalent in their ability to support increased rates of MPS. A recent study confirmed that a blend of plant proteins at a large dose of 30 g resulted in similar MPS as 30g of milk protein in young men. However, the impact of a unique plant-derived protein blend on MPS in older individuals is yet to be determined. Therefore, the purpose of this study is to address that knowledge gap by assessing the skeletal muscle anabolic potential of a plant-based protein blend (i.e., corn and pea) on rates of MPS, with or without additive exercise in older men and women.

ELIGIBILITY:
Inclusion Criteria:

* Older (60-80 y) men and women
* Be in good general health
* Non-smoking
* Recreationally active but not meet Canada's Physical Activity Guidelines (150 min of moderate-intensity exercise/week)
* Have a body mass index (BMI) between 18.5-30 kg/m2 (inclusive)
* Willing and able to provide informed consent (speaks and understands English)

Exclusion Criteria:

* Use of tobacco or related products
* Use assistive walking devices (e.g., cane or walker)
* Any concurrent medical, orthopedic, or psychiatric condition that, in the opinion of the investigator, would compromise his/her ability to comply with the study requirements
* History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years
* Significant orthopedic, cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, metabolic/endocrine, neuromuscular or bone wasting disorders
* Any cachexia-related condition (e.g., relating to cancer, tuberculosis or human immunodeficiency virus infection and acquired immune deficiency syndrome) or any genetic muscle diseases or disorders
* History of statin myalgia
* Current illnesses which could interfere with the study (e.g., prolonged severe diarrhea, regurgitation, difficulty swallowing)
* Excessive alcohol consumption (>21 units/week)
* History of bleeding diathesis, platelet or coagulation disorders, or antiplatelet/anticoagulation therapy (up to 81mg of baby aspirin per day taken as a prophylactic is permitted).
* Routine/daily usage of non-steroidal anti-inflammatory drugs (NSAIDS, prescription use or daily use of over-the-counter medication), use of corticosteroids, testosterone replacement therapy (ingestion, injection, or transdermal), any anabolic steroid, creatine, whey protein supplements, casein or branched-chain amino acids (BCAAs) within 45 days prior to screening.
* A history of falls determined by a score >25 on the Falls Efficacy Scale-International (FES-I).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Muscle protein synthesis rate | Over 5 hours after intervention
  The rate of amino acids incorporation into skeletal muscle protein

SECONDARY OUTCOMES:
Plasma amino acid concentration | Over 5 hours after intervention
  Amino acid content in plasma after ingestion of the supplements
Muscle anabolic protein signaling | At pre and 5 hours after intervention
  Protein signaling changes in skeletal muscle tissue
Plasma glucose | Over 5 hours after intervention
  Glucose content in plasma
Plasma insulin | Over 5 hours after intervention
  Insulin content in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, Ph.D., Principal Investigator — McMaster University
Locations (1):
- Ivor Wynne Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No